CLINICAL TRIAL: NCT07270068
Title: Remission of Diabetes With Lifestyle Intervention for Malaysian Type 2 Diabetes Mellitus Patients (ReDiaL-MY) - an Open Label, Randomised Controlled Study
Brief Title: Remission of Diabetes With Lifestyle Intervention for Malaysian Patients
Acronym: ReDiaL-MY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Winnie Chee Siew Swee (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Sponsor-Investigator, Winnie Chee Siew Swee, Director of Institute for Research, Development and Innovation (IRDI), IMU University
Organization: IMU University, Malaysia (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ReDiaL-MY
Record Dates: First submitted 2025-11-21; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Type 2 diabetes mellitus; Remission; Malaysia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a randomised wait-list-controlled trial, that consists of :
  i) a randomised clinical trial phase (6 months) and ii) an observational follow-up phase (6 months)
  Participants will be randomised either to commence the intervention immediately after randomisation (intervention group), or to continue usual management of T2DM for six months, prior to starting the intervention (wait-list control group).
  Thereafter, the intervention group would enter the weight maintenance phase for another 6 months. The wait-list control would be offered the intervention for 6 months and follow-up on the weight maintenance, similar to the intervention group.
  This study design will provide comparisons between groups during the randomised phase of 6 months, and observational data in an enlarged cohort (wait-list control + intervention) on weight maintenance phase for and additional 6 month.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The Intervention group will undergo total diet replacement (TDR) phase for 8-12 weeks of followed by food reintroduction (12-16 weeks). After the RCT phase (up to 16 weeks), the intervention group enters a weight maintenance period for 24 weeks.
  The participant will be given 4 servings Diabetes-specific formula (DSF) of Glucerna® Control Vanilla Flavour or 3 servings of DSF with additional ~300 kcal low calorie low glycaemic index portion-controlled meal for daily consumption within a minimum of 8 weeks to a maximum of 12 weeks during the TDR phase. In the food reintroduction phase, there will be a gradual replacement of the DSF with low calorie low glycemic index portion-controlled meals. While in the weight maintenance phase, participants will be offered the use of 1 DSF a day as part of their healthy diet plan (1200 - 1500 kcal/day).
  Interventions: Dietary Supplement: Total Diet Replacement
- Wait List Control (Active Comparator): The wait-list control group will follow the usual care consisting of conventional diet plan and routine physician care for the initial 24 weeks of intervention parallel to the Intervention group. Upon completion of the 24 weeks of the intervention group, the wait-list control group will crossover to receive the similar intervention and observation plans as per the intervention group.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Dietary Supplement: Total Diet Replacement — Total Diet Replacement (TDR) Phase (8-12weeks), followed by Food reintroduction phase (12-16 weeks) (8 to 12 weeks = 4 months)
  Arms: Intervention group
Behavioral: Standard of Care — conventional diet plan and routine physician care
  Arms: Wait List Control

SUMMARY:
This study aims to evaluate the effectiveness of structured lifestyle intervention to induce remission of Type 2 Diabetes Mellitus (T2DM) among Malaysian adults. The study will also assess the feasibility of implementing this intervention within Malaysian primary and specialist care settings. The study will also examine the economic impact of the TDR intervention through a cost-effectiveness analysis conducted from a societal perspective.

Researchers will compare intensive lifestyle intervention to the usual clinical care.

It is hypothesised that Malaysian adults with T2DM who receive the structured lifestyle intervention will demonstrate a significantly higher rate of diabetes remission compared to those receiving usual care. Furthermore, participants in the intervention group are expected to achieve greater mean weight loss, with a higher proportion attaining a sustained weight loss of at least 10 kilograms, relative to the usual care group. The lifestyle intervention is also anticipated to result in superior glycaemic control, as measured by reductions in glycated haemoglobin (HbA1c), and to be more cost-effective in achieving diabetes remission and reducing long-term healthcare utilization.

DETAILED DESCRIPTION:
Malaysia is facing an epidemic of diabetes and despite public health efforts to increase awareness, screening and prevention, there is a continued rise in the prevalence of diabetes and its complications. A lifestyle approach for diabetes remission may be a solution to curb further rise in diabetes complications and be cost-effective.

Little is known about the transferability of diabetes remission lifestyle intervention into Malaysian primary care settings. This knowledge is important to understand whether DiRECT is feasible, actionable and acceptable to patients, clinicians and primary care settings given the original trial was developed overseas. Furthermore, local data on the economic burden of diabetes and the potential savings from remission are urgently needed to support evidence-based policymaking. This study will therefore include an economic evaluation using a cost-of-illness approach with a prevalence-based model, incorporating both direct and indirect costs from the societal perspective. In addition, the results from this proposed study will be important to see how we can increase acceptability of this approach in Malaysia and curb a disabling disease that is rapidly rising in Malaysia.

This study is a randomised, wait-list-controlled, dual-phase trial designed to evaluate the efficacy and cost-effectiveness of a structured lifestyle intervention for inducing remission of Type 2 Diabetes Mellitus (T2DM) in Malaysian adults. The protocol integrates a rigorous clinical trial framework with a comprehensive economic evaluation from a societal perspective.

The trial employs a randomised wait-list-controlled design, comprising two distinct phases:

1. Randomised Controlled Trial (RCT) Phase: Eligible participants are randomised in a 1:1 ratio, using a computer-generated sequence via an online software (Sealed Envelope), to either the immediate intervention group or a wait-list control group. The structured intervention is undergo 12 weeks of total diet replacement course, followed by food reintroduction (12 weeks). The wait-list group will receive standard of care for the primary endpoint assessment at 24 weeks.
2. Observational Follow-up Phase: Following the RCT phase, the intervention group enters a weight maintenance period. The wait-list control group crosses over to receive the identical structured intervention for 24 weeks. This phase provides longitudinal data on weight maintenance and diabetes remission sustainability in an enlarged cohort for up to 12 months.

Definition of three sequential phases are:

Total Diet Replacement (TDR) Phase (8-12 weeks) aims to rapid weight loss, targeting a 15% reduction from baseline body weight. This is achieved through a hypocaloric regimen of approximately 800-850 kcal per day. Support during this phase includes two face-to-face appointments in the first month, followed by monthly face-to-face/virtual contacts and bi-weekly phone calls with a study dietitian.

Food Reintroduction Phase (12-16 weeks) facilitates a structured transition from TDR to a solid-food-based diet for weight maintenance. Using a stepped protocol, the DSF is gradually replaced over several weeks with low-calorie, low-glycaemic index meals, increasing total daily energy intake from 1000 kcal to 1400 kcal. Participants are subsequently advised to titrate their intake by 200 kcal increments until a stable weight is achieved. Dietary counseling utilising motivational interviewing techniques is introduced to reinforce behavioural changes. Support includes two face-to-face appointments in the first month, followed by monthly face-to-face/virtual contacts and bi-weekly phone calls.

Weight Maintenance Phase (24 weeks) The focus shifts to sustaining lifestyle changes and preventing weight regain. Participants follow a healthy diet plan (1200-1500 kcal/day) and are offered one DSF serving daily as a dietary component. Physical activity of at least 150 minutes per week is recommended. Support is maintained through six face-to-face or virtual contacts with the dietitian.

Integrated Medical Management and Relapse Protocol will be chaired by certified Medical Officers. A critical and technically detailed component of the protocol is the systematic management of concomitant medications and weight regain. The medical is responsible and cover the below aspect.

1. Medication Withdrawal: Upon TDR initiation, all oral hypoglycaemic agents (OHA), antihypertensives, and diuretics are withdrawn to mitigate risks of hypoglycaemia and hypotension, with reinstatement protocols based on strict systolic blood pressure (BP) and glycaemic thresholds.
2. Hypertension Management: Antihypertensives are reintroduced in a defined sequence (ACE inhibitors → ARBs → Thiazides → etc.) if systolic BP exceeds 165 mmHg in the first two weeks, or >140 mmHg thereafter, with weekly dose titrations.
3. Glycaemic Management Protocol: If troublesome hyperglycaemic symptoms or random capillary glucose >20 mmol/L persist after two weeks of TDR, glucose-lowering medications are reintroduced in a stepped manner
4. Relapse Management: A "rescue plan" is activated for participant have trouble to reduce weight and blood glucose. Nevertheless, biomarkers rebound to a unsafe level. Medical team might consider revert the participants back to standard of care and reintroduction medications for controlling diabetes.

monitored via 3-day food records and daily DSF consumption logs, with compliance calculated as a percentage of actual versus expected intake.

A nested qualitative study uses semi-structured, theory-domain interviews to explore barriers and facilitators to diabetes remission. Patients are interviewed at four timepoints (Baseline, 12 weeks, 6 months, and 12 months). Additionally, a purposive sample of 10-15 healthcare professionals involved in intervention delivery will be interviewed to assess implementation barriers and facilitators.

Participants are closely monitored for Adverse Events (AEs). Blood pressure, postural symptoms, and capillary blood glucose will be All AEs are recorded and reported, with Serious AEs reported to the Ethics Committee within 48 hours. A clinical trial insurance will be secured for all participants.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed diabetes for a duration of < 3 years (diagnosis based on 2 recorded diagnostic-level tests, HbA1C and/or blood glucose)
2. Body mass index (BMI) > 25 kg/m2
3. HbA1C level above > 6.5% to 9% as per the last routine clinical check within 6 months
4. Currently being treated with one or more oral glucose lowering drugs

Exclusion Criteria:

1. Type 1 DM
2. Type 2 DM on basal or multiple insulin injections
3. Recent routine HbA1C of > 9%
4. Patients who in the past 6 months have weight loss exceeding 5 kg (such individuals may have difficulty losing additional weight)
5. Recent (last 12 weeks) or current use of medications/meal replacements for weight loss
6. Alcoholism or any substance abuse
7. History of bariatric surgery, small bowel resection, or extensive bowel resection
8. Chronic treatment with systemic corticosteroids. Use of hormone replacement therapy or oral contraceptives will not lead to exclusion
9. Severe hypertension on multiple drugs treatment
10. Currently pregnant or nursing and planning to get pregnant
11. Requiring hospitalization for depression or are on antipsychotic medications
12. Cancer requiring treatment for the past 5 years, except of non-melanoma skin cancers or cancers that have been clearly cured
13. HIV- positive (self-report) due to effects or weight and body composition of HIV and medications treating HIV
14. Cardiovascular disease (heart attack or procedure within past 3 months or participation in cardiac rehabilitation program within last 3 months, stroke or history/ treatment for transient ischemic attacks in the past 3 months, or documented history of pulmonary embolus for the past 6 months)
15. Renal disease - eGFR < 60 ml/min (based MDRD) or currently receiving dialysis
16. Proliferative retinopathy and other severe diabetes complications
17. Diagnosed eating disorder or purging

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving diabetes remission | 6 months
  Diabetes remission defined as HbA1C ≤ 6.5% or ≤48 mmol/mol and no diabetes medication required.

SECONDARY OUTCOMES:
Proportion of patients maintaining diabetes remission | 12 months
  Diabetes remission defined as HbA1C ≤ 6.5% or ≤48 mmol/mol and no diabetes medication required.
Weight loss | 12 weeks, 6 months and 12 months
  Changes of Weight (kg)
Insulin Resistance (HOMA-IR) | 12 weeks, 6 months and 12 months
  Calculate the body's tissues respond to insulin to take up glucose. [Fasting insulin (U/ml) x fasting plasma glucose (mg/dl)] / 405
Pancreatic β-cell function (HOMA-β) | 12 weeks, 6 months and 12 months
  Calculate the functions of pancreas in producing insulin. [20 x fasting insulin (U/ml)] / [fasting plasma glucose (mg/dl) - 63]

OTHER OUTCOMES:
Physical Functions | 12 weeks, 6 months and 12 months
  Measure the time need to complete a 5-times sit-to-stand test and/or 6-meters walk test
Muscle Strength | 12 weeks, 6 months and 12 months
  Changes of kilograms-force (using dynamometer)
Monitoring Biomarker | 12 weeks, 6 months and 12 months
  Changes of kidney and liver functions
Cost-effectiveness | 6 months and 12 months
  Direct and indirect medical expenses from societal perspective

CONTACTS AND LOCATIONS:
Overall Officials: Winnie Siew Swee Chee, PhD, Principal Investigator — IMU University
Locations (2):
- Malaysia (2):
  - Klinik Kesihatan Seremban, Seremban, Negeri Sembilam
  - Hospital Putrajaya, Kuala Lumpur, Putrajaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor R. Aetiology of type 2 diabetes: an experimental medicine odyssey. Diabetologia. 2025 Jul;68(7):1375-1389. doi: 10.1007/s00125-025-06428-0. Epub 2025 May 2. PMID 40316731
- [Background] Sattar N, Welsh P, Leslie WS, Thom G, McCombie L, Brosnahan N, Richardson J, Gill JMR, Crawford L, Lean MEJ. Dietary weight-management for type 2 diabetes remissions in South Asians: the South Asian diabetes remission randomised trial for proof-of-concept and feasibility (STANDby). Lancet Reg Health Southeast Asia. 2023 Feb;9:100111. doi: 10.1016/j.lansea.2022.100111. PMID 36777452
- [Background] Lean MEJ, Leslie WS, Barnes AC, Brosnahan N, Thom G, McCombie L, Peters C, Zhyzhneuskaya S, Al-Mrabeh A, Hollingsworth KG, Rodrigues AM, Rehackova L, Adamson AJ, Sniehotta FF, Mathers JC, Ross HM, McIlvenna Y, Welsh P, Kean S, Ford I, McConnachie A, Messow CM, Sattar N, Taylor R. Durability of a primary care-led weight-management intervention for remission of type 2 diabetes: 2-year results of the DiRECT open-label, cluster-randomised trial. Lancet Diabetes Endocrinol. 2019 May;7(5):344-355. doi: 10.1016/S2213-8587(19)30068-3. Epub 2019 Mar 6. PMID 30852132

DOCUMENTS (1):
  • Informed Consent Form (2025-05-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT07270068/ICF_000.pdf